CLINICAL TRIAL: NCT05864365
Title: An Open-Label Biomarker Study of ATH434 in Multiple System Atrophy
Brief Title: A Biomarker Study of ATH434 in Participants With MSA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alterity Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATH434-202
Record Dates: First submitted 2023-05-09; First posted 2023-05-18 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Multiple System Atrophy
Keywords: Multiple System Atrophy; ATH434; Neurodegenerative disease; Shy-Drager Syndrome; Movement disorders; Autonomic dysfunction; Synucleinopathies; Atypical parkinsonism; Biomarkers
MeSH Terms: conditions — Multiple System Atrophy; Neurodegenerative Diseases; Shy-Drager Syndrome; Movement Disorders; Primary Dysautonomias; Synucleinopathies | interventions — ATH434

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- ATH434 (Experimental)
  Interventions: Drug: ATH434

INTERVENTIONS:
Drug: ATH434 — ATH434 taken by mouth two times per day

SUMMARY:
This study will assess the safety and efficacy of ATH434 in participants with a clinical diagnosis of Multiple System Atrophy

ELIGIBILITY:
Inclusion Criteria:

1. Participant has clinical features of parkinsonism.
2. Participant has evidence of orthostatic hypotension and/or bladder dysfunction.
3. Participant has ataxia and/or pyramidal signs on neurological examination.
4. Participant has biomarker evidence of MSA in biologic fluid and on MRI.

Exclusion Criteria:

1. Participant is unable to swallow study drug.
2. Participant is unable to attend study visits or complete study procedures.
3. Participant has structural brain abnormality on MRI.
4. Participant has any significant neurological disorder other than MSA.
5. Participant has an unstable medical or psychiatric illness.
6. Participant has a contraindication to, or is unable to tolerate, MRI or lumbar puncture.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-05-23 (Actual); Primary Completion 2025-02-26 (Actual); Study Completion 2025-02-26 (Actual)

PRIMARY OUTCOMES:
Change in brain volume as measured by MRI | Change from Baseline to Week 52

SECONDARY OUTCOMES:
Change in iron content in substantia nigra as measured by MRI | Change from Baseline to Week 52
Change in Unified MSA Rating Scale (UMSARS) Score | Change from Baseline to Week 52
Change in Patient Global Impression of Change (PGI-C) | Change from Baseline to Week 52
Change in Clinical Global Impression of Change (CGI-C) | Change from Baseline to Week 52
Change in Neurofilament Light Chain Levels | Change from Baseline to Week 52

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No